CLINICAL TRIAL: NCT01091766
Title: Sensitivity of Electrocardiogram on Detection of Three Different Intravascular Applied Test Doses of Bupivacaine and Epinephrine: a Study in Children of Different Age
Brief Title: Sensitivity of ECG on Detection of Three Different Intravascular Applied Test Doses of Bupivacaine and Epinephrine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Children's Hospital, Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: StV 25/09
Record Dates: First submitted 2010-03-22; First posted 2010-03-24 (Estimated); Last update posted 2012-07-24 (Estimated); Status verified 2012-07

CONDITIONS: Anaesthesia; Toxicity
Keywords: local anaesthetics toxicity; heart arrhythmia; heart rate; heart conduction; regional anaesthesia; paediatric anaesthesia; cardio-vascular system; prevention
MeSH Terms: conditions — Arrhythmias, Cardiac

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- bupivacaine (Active Comparator): test solution consists of bupivacaine 0.125%
  Interventions: Drug: intravenous injection of test solution
- bupivacaine+epinephrine (Active Comparator): test solution consists of bupivacaine 0.125% with epinephrine 1:200000
  Interventions: Drug: intravenous injection of test solution
- epinephrine (Active Comparator): test solution consists of epinephrine 1:200000
  Interventions: Drug: intravenous injection of test solution

INTERVENTIONS:
Drug: intravenous injection of test solution — test dose consists of 0.2 ml/kg body weight test solution of the assigned drug
  Arms: bupivacaine
Drug: intravenous injection of test solution — test dose consists of 0.2 ml/kg body weight test solution of the assigned drug
  Arms: bupivacaine+epinephrine
Drug: intravenous injection of test solution — test dose consists of 0.2 ml/kg body weight test solution of the assigned drug
  Arms: epinephrine

SUMMARY:
The purpose of this prospective randomised study is to investigate electrocardiographic alterations after intravascular injection of three different test solutions of bupivacaine and epinephrine in anaesthetised children up to 16 years of age.

ELIGIBILITY:
Inclusion Criteria:

* Age 0 to 16
* healthy
* parental consent

Exclusion Criteria:

* ASA >1
* allergy against local anaesthetics

Ages: 1 Day to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 150 (Actual)
Dates: Start 2010-03; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
T-wave elevation in the ECG after intravenous administration of the test solution | 2 minutes
  0.2 ml/kg test solution (bupivacaine or bupivacaine+epinephrine or epinephrine) is intravenously injected. The ECG is recorded over 2 minutes, printed and analysed later on regarding alterations of T-wave.

SECONDARY OUTCOMES:
Alteration in heart rate caused by intravenous injection of the test solution | 2 minutes
  0.2 ml/kg test solution (bupivacaine or bupivacaine+epinephrine or epinephrine) is intravenously injected. The ECG is recorded over 2 minutes, printed and analysed later on regarding alterations in heart rate.

CONTACTS AND LOCATIONS:
Overall Officials: Markus Weiss, Prof, Principal Investigator — University Childrens Hospital Zurich, Anesthesiology
Locations (1):
- University Children's Hospital, Anesthesiology, Zurich, Switzerland

REFERENCES:
- [Result] Mauch J, Kutter AP, Madjdpour C, Koepfer N, Frotzler A, Bettschart-Wolfensberger R, Weiss M. Electrocardiographic alterations during intravascular application of three different test doses of bupivacaine and epinephrine: experimental study in neonatal pigs. Br J Anaesth. 2010 Jan;104(1):94-7. doi: 10.1093/bja/aep313. PMID 19915187